CLINICAL TRIAL: NCT00426075
Title: Full-Leg vs Below-Knee Elastic Stockings for Prevention of the Post-Thrombotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Paolo Prandoni, Department of Medical and Surgical Sciences, University of Padua
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11/98
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis of the lower extremities
MeSH Terms: conditions — Venous Thrombosis | interventions — Stockings, Compression

INTERVENTIONS:
Device: Elastic stockings

SUMMARY:
Prospective controlled randomized clinical trial. Consecutive patients with acute proximal deep vein thrombosis of the lower extremities, with or without contemporary manifestations of pulmonary embolism, are randomized to receive either a below-knee or a full-leg graduated compression (30-40 mm Hg at the ankle) elastic stocking for prevention of the post-thrombotic syndrome (PTS). All patients are followed up to three years to assess the development of the PTS, defined according to a validated clinical score (the Villalta scale). The rate of PTS is compared between the two study groups. In addition, there is an assessment of patients' compliance and tolerability of the two different devices.

ELIGIBILITY:
Inclusion Criteria:

* First episode of proximal deep vein thrombosis, as shown by compression ultrasound

Exclusion Criteria:

* Previous ipsilateral deep vein thrombosis
* Preexisting chronic venous insufficiency
* Bilateral deep vein thrombosis
* Life expectancy lower than 1 year
* Severe arteriopathy of the lower limbs
* Known allergy to elastic stockings
* Lack of written informed consensus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-01; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Prandoni, MD, PhD, Principal Investigator — Department of Medical and Surgical Sciences, University of Padua, Italy
Locations (1):
- Department of Medical and Surgical Sciences, 2nd Chair of Internal Medicine, University of Padua, Padua, Padua, Italy

REFERENCES:
- [Derived] Prandoni P, Noventa F, Quintavalla R, Bova C, Cosmi B, Siragusa S, Bucherini E, Astorri F, Cuppini S, Dalla Valle F, Lensing AW, Prins MH, Villalta S; Canano Investigators. Thigh-length versus below-knee compression elastic stockings for prevention of the postthrombotic syndrome in patients with proximal-venous thrombosis: a randomized trial. Blood. 2012 Feb 9;119(6):1561-5. doi: 10.1182/blood-2011-11-391961. Epub 2011 Dec 16. PMID 22180438